CLINICAL TRIAL: NCT03318055
Title: Evaluating Perioperative Interventions to Improve Patient Outcomes (EPIC-1) Study
Brief Title: Prevalence of Hyperglycemia and Anaemia in Elective Surgical Patients
Acronym: EPIC-1
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Professor, University of Cape Town
Other Study IDs: EPIC1
Record Dates: First submitted 2017-10-06; First posted 2017-10-23 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Anemia, Iron Deficiency; Hyperglycemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group study: The study population will include patients presenting for elective surgery, who fulfil the inclusion criteria of all surgical disciplines undergoing elective surgery period during the period of the study.
  Inclusion Criteria:
  > 18 years of age Non-cardiac patients Non-obstetric patients Patients receiving general, neuraxial, regional or local/topical anaesthesia for elective surgical intervention

SUMMARY:
The study is a prospective, observational study of adult, non-cardiac, non-obstetric, elective surgical patients conducted over a period of one week. This large-scale clinical audit aims to assess the incidence rates of anaemia and hyperglycaemia amongst elective surgical patients in the Western Cape. A study such as this is essential in the assessment of the incidence rates of abnormal fasting blood glucose levels and reduce the risk of perioperative complications for patients. Preoperative anaemia is a modifiable risk factor and should be identified early and treated appropriately to improve patient outcomes.

DETAILED DESCRIPTION:
Globally, one third of patients presenting for surgery will be anaemic, according to the WHO criteria. Preoperative anaemia is considered an independent risk factor for poorer patient outcomes, with increases in morbidity and mortality as well as prolonged length of hospital stay. However, the importance of this finding in the preoperative period is often overlooked and not corrected prior to surgery. The leading cause of preoperative anaemia is iron deficiency. Iron deficiency anaemia is common in developing countries and results mostly from nutritional deficiency. Poorly controlled Diabetes Mellitus (DM) is known to have an adverse effect on perioperative clinical outcomes, with an extended length of hospital stay and increased morbidity and mortality. Preoperative identification of patients with DM, provides a potential opportunity to reduce the risk of adverse surgical outcomes. Early identification of such patients could facilitate timely intervention and arrangement of appropriate perioperative and long-term follow-up. Studies have demonstrated that an elevated HbA1c (indicative of poor glycaemic control in the months preceding surgery) correlates with increased perioperative risk in known diabetics. On the day of surgery, before induction of anaesthesia, all patients will have a finger prick blood glucose level done by point of care glucometry, if there is no documented fasting blood glucose value in their ward file. In patients of unknown diabetic status, should the preoperative value be >7 mmol/l, blood will be drawn when IV access is established, for HbA1C measurement. In known diabetics, a sample will be taken for HbA1C, regardless of the preoperative fasting blood glucose level, unless there is an HbA1C measurement in the previous 3 months. However, should the patient management have been modified based on the HbA1C result, a repeat HbA1C measurement would be performed

All patients will be assessed as part of the routine preoperative evaluation. Informed consent will be obtained by the anaesthetist from eligible patients who agree to participate in the study. On the day of surgery, prior to induction of anaesthesia the patients will receive a finger prick Hemoglobin (Hb) if they have not had a Hb result documented within the last 3 months. If the results meet the WHO criteria for anemia, a blood specimen will be collected when inserting the IV line. The blood specimen will be sent for Haemoglobin, mean cell volume, ferritin and transferrin saturation (TSAT) testing. All patients diagnosed with anemia will receive a patient information leaflet. They will also be referred to their local clinics or general practitioner for further evaluation and appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Adult, non-cardiac, non-obstetric, elective surgical patients

Exclusion Criteria:

* Obstetric, emergency and cardiac patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises all adult non-cardiac, non-obstetric patients presenting for elective surgery over a period of one week at following sites: Groote Schuur -, Somerset -, Paarl -, Victoria -, Mitchell's Plain - and George Hospital.
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of diagnosis of diabetes and anaemia | Day of surgery
  Proportion of patients with diagnosis of diabetes and anaemia

SECONDARY OUTCOMES:
HbA1C level | Day of surgery
  Assessment of diabetic control
Transferrin saturation | Day of surgery
  Diagnosis of iron deficiency anaemia
Serum ferritin | Day of surgery
  Diagnosis of iron deficiency anaemia

CONTACTS AND LOCATIONS:
Overall Officials: Netjhardt Marcin, MBChB, FCA, Principal Investigator — University of Cape Town; Francois Roodt, MBChB, FCA, Principal Investigator — University of Cape Town
Locations (6):
- South Africa (6):
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Mitchells Plain Hospital, Cape Town, Western Cape
  - Somerset Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - George Hospital, George, Western Cape
  - Paarl Hospital, Paarl, Western Cape

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03318055/Prot_000.pdf